CLINICAL TRIAL: NCT01411462
Title: Vascular Imaging Balloon Catheter-assisted Drug-eluting Balloon Angioplasty Prospective Registry
Brief Title: VIBE-assisted DEB Registry
Acronym: VIBER
Status: Withdrawn | Type: Observational
Why Stopped: Funding issues
Sponsor: Ospedale Santa Maria Goretti (Other)
Responsible Party: Principal Investigator, Gregory Sgueglia, MD, Dr, Ospedale Santa Maria Goretti
Other Study IDs: SMG-007
Record Dates: First submitted 2011-08-03; First posted 2011-08-08 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- VIBE-DEB
  Interventions: Device: VIBE + drug-eluting balloon

INTERVENTIONS:
Device: VIBE + drug-eluting balloon — VIBE before and after durg-eluting balloon angioplasty

SUMMARY:
VIBER aims at assessing angiographic outcome of drug-eluting balloon angioplasty assisted by the Vascular Imaging Balloon Catheter (VIBE, Volcano, San Diego, CA) device, which integrates a predilation catheter with electronic intravascular ultrasound capabilities.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* De novo native vessel lesion
* RVD 2.5 - 4 mm Limited compliance with >3 month DAPT

Exclusion Criteria:

* LMCA

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with symptomatic coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-08 (Estimated); Primary Completion 2011-10 (Estimated); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Binary restenosis | 6 months
  Number of patients with a diameter stenosis >50% assessed by quantitative coronary angiography

SECONDARY OUTCOMES:
Procedural success | 1 day
  Number of patients with both post-procedure diameter stenosis <20% assessed by quantitative coronary angiography and TIMI 3 flow
Major adverse cardiac events | 6 months
  Number of patients with one of the following events: cardiac death, non-fatal myocardial infarction, target lesion revascularization

CONTACTS AND LOCATIONS:
Locations (1):
- S.M. Goretti, Latina, Italy